CLINICAL TRIAL: NCT04859829
Title: Autoimmune Gastrointestinal Dysmotility: Symptoms, Pathogenesis and Treatment
Status: Terminated | Type: Observational
Why Stopped: PI moved to another institution and closed study.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00087869
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2022-03

CONDITIONS: Dysmotility Syndrome; Autoimmunity
MeSH Terms: conditions — Ciliary Motility Disorders; Autoimmune Diseases | interventions — Immunoglobulins, Intravenous; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with autoimmune dysmotility receiving IVIG infusions
  Interventions: Other: Current Intravenous Immunoglobulin (IVIG) treatment
- Patients with autoimmune dysmotility without IVIG infusions
  Interventions: Other: No Intravenous Immunoglobulin (IVIG) treatment

INTERVENTIONS:
Other: Current Intravenous Immunoglobulin (IVIG) treatment — Questionnaires every two months for patients with a diagnosis of autoimmune dysmotility that are receiving Intravenous Immunoglobulin (IVIG) treatment.
  Groups: Patients with autoimmune dysmotility receiving IVIG infusions
Other: No Intravenous Immunoglobulin (IVIG) treatment — Questionnaires every two months for patients with a diagnosis of autoimmune dismotility that are not receiving Intravenous Immunoglobulin (IVIG) treatment.
  Groups: Patients with autoimmune dysmotility without IVIG infusions

SUMMARY:
Autoimmune gastrointestinal dysmotility syndromes are poorly understood, and often difficult to treat because the underlying pathogenesis is unclear. Refractory symptoms result in an impaired quality of life. The presence of positive serum autoantibodies to peripheral nervous system gangliosides and glycoproteins is suggestive of a possible mechanism. Immunomodulator treatments have shown benefit in case reports and case series but standardized data for treatment response is lacking. Therefore, our primary aims are to further characterize this syndrome in terms of symptoms, laboratory testing, pathology, and assess treatment response of immunomodulator therapy. Our research plan involves identifying this subset of patients with autoimmune gastrointestinal dysmotility and dysautonomia, and studying them as they are managed by their gastroenterologists.The study team will administer symptom-based questionnaires in a systematic manner to assess the clinical trajectory of this population and treatment response. The investigators will also analyze laboratory values (antibody titers, tilt testing, inflammatory markers) and study pathology specimens (enteric and skin biopsies) obtained from this cohort to gain a deeper understanding of the pathogenesis of their disease.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, Aged>15
* Evidence of enteric dysmotility with documented abnormality on objective testing which may include high resolution esophageal manometry, gastric emptying scintigraphy, SmartPill Wireless Motility Capsule, Sitz marker studies, antroduodenal manometry or anorectal manometry.
* English proficiency and literacy sufficient to sign consent form and fill out questionnaires.
* Previous Mayo paraneoplastic panel testing.
* Referring gastroenterologist has recommended intravenous immunoglobulin (IVIg) therapy.

Exclusion Criteria:

* Non-autoimmune causes of enteric dysmotility (diabetes, adrenal insufficiency, Parkinson's, thyroid, electrolytes, drugs, malignancy).
* Pregnancy as documented in EPIC with serum or urine Human chorionic gonadotropin (hCG) testing

  * If participants believe that they are pregnant, they will need to notify a study physician who will order a serum or urine hCG test for pregnancy within EPIC and remove them from the study if the test results come back positive.
* Previous treatment with IVIg.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with autoimmune autonomic ganglionopathy (AAG) or autoimmune autonomic neuropathy. Postural orthostatic tachycardia syndrome (POTS) and gastrointestinal (GI) dysmotility.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Change in upper gastrointestinal symptom severity as assessed by the Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index | Every two months up to 2 years.
  The Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index (PAGI-SYM) is composed of 20 items and 6 sub-scales: heartburn/regurgitation (7 items), nausea/vomiting (3 items), postprandial fullness/early satiety (4 items), bloating (2 items), upper abdominal pain (2 items), and lower abdominal pain (2 items). Sub-scale scores are calculated by averaging across items comprising the sub-scale; scores vary from 0 (none or absent) to 5 (very severe).

SECONDARY OUTCOMES:
Change in Quality of Life as assessed by the Patient Assessment of Upper Gastrointestinal Disorders-Quality of Life scale | Every two months up to 2 years.
  The effect of Autoimmune Dysmotility symptoms on quality of life assessed by the Patient Assessment of Upper Gastrointestinal Disorders-Quality of Life (PAGI-QoL). The PAGI-QOL instrument consists of 30 items, each with response options based on a 6-point scale and with a recall period of the previous 2 weeks. The items are grouped into 5 dimensions: Daily Activities, Clothing, Diet and Food Habits, Relationship and Psychological Well-being and Distress. A score per dimension as well as a total score can be calculated. The PAGI-QOL scores range from 0 (lowest QoL) to 5 (highest QoL).

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj J Pasricha, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Pasricha PJ, McKnight M, Villatoro L, Barahona G, Brinker J, Hui K, Polydefkis M, Burns R, McMahan ZH, Gould N, Goodman B, Hentz J, Treisman G. Joint Hypermobility, Autonomic Dysfunction, Gastrointestinal Dysfunction, and Autoimmune Markers: Clinical Associations and Response to Intravenous Immunoglobulin Therapy. Am J Gastroenterol. 2024 Nov 1;119(11):2298-2306. doi: 10.14309/ajg.0000000000002910. Epub 2024 Jun 24. PMID 38912927